CLINICAL TRIAL: NCT01166100
Title: A Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover Bioequivalence Study of Fluoxetine Hydrochloride Delayed-Release Capsules 90 mg of Dr. Reddy's and Prozac®Weekly 90 mg DR Capsules of Eli Lilly and Company, USA in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Fluoxetine Hydrochloride Delayed-Release Capsules, 90 mg of Dr. Reddy's Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Mr. M.S. Mohan / Vice President (Research and Development), Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 587/05
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Fluoxetine Hydrochloride
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine Hydrochloride (Experimental): Fluoxetine Hydrochloride Delayed-Release Capsules, 90 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Fluoxetine Hydrochloride
- Prozac ® weekly TM (Active Comparator): Prozac ® weekly 90 mg delayed release capsules of Eli Lilly and company
  Interventions: Drug: Fluoxetine Hydrochloride

INTERVENTIONS:
Drug: Fluoxetine Hydrochloride — Fluoxetine Hydrocloride Delayed Release Capsules, 90 mg of Dr. Reddy's Laboratories.
  Other Names: Prozac ® weekly 90 mg Delayed-Release Capsules

SUMMARY:
The purpose of this study is to asses the bioequivalence study of Fluoxetine Hydrochloride Delayed-Release Capsules, 90 mg and Prozac ® weekly under fasting conditions.

DETAILED DESCRIPTION:
A randomized, open label, two treatment, two period, two sequence, single dose, crossover bioequivalence study of Fluoxetine Hydrochloride delayed release capsules 90 mg of Dr. Reddy's laboratories limited, Generics, India and Prozac®weekly 90 mg delayed release capsules of Eli Lilly and company, USA in healthy adult human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects between 18-50 years of age (inclusive), weighing as per the standard height and weight chart of Life Insurance Corporation of India (11 Underweight and Overweight Min. & Max. Chart).
* Subjects who have no evidence of underlying disease during screening medical history and whose physical examination is performed within 21 days prior to commencement of the study.
* Subjects whose screening laboratory values are within normal limits or considered by the physician/Principal Investigator to be of no clinical significance.
* Informed consent given in written form according to section 11.3 of the protocol.
* Female Subjects

  * of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies,diaphragm, intrauterine device, or abstinence.
  * postmenopausal for at least I year.
  * surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

* Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
* Alcohol dependence, Alcohol abuse, i.e., regular use of more than 2 units of alcohol or 10 units per week or a history of alcoholism (one unit of alcohol equals 1/2 1 of beer 200 ml wine or 50 ml (of spirits) within last 6 months or recovered alcoholics , or drug abuse within past 1 year.
* Moderate to heavy smoking (> 10 cigarettes/day) or consumption of tobacco products.
* History of difficulty in swallowing capsules.
* Clinically significant illness within 4 weeks before the start of the study.
* Asthma, urticaria or other allergic type reactions after taking any medication.
* Positive urine drug screening, Human Immunodeficiency Virus, Hepatitis B & C tests.
* Any history of hypersensitivity to fluoxetine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-02; Primary Completion 2006-03 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. James John, MBBS, MD, Principal Investigator — Lotus Labs Private Limited
Locations (1):
- Lotus Labs Private Limited, Mylapore, Chennai, India